CLINICAL TRIAL: NCT00841711
Title: Transitions: Linkages From Jail to Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0711003262; H97HA08541
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: HIV; Substance Abuse; HIV Infections
Keywords: HIV; AIDS; Buprenorphine; Intensive Case Management; Money Management; Rapid Testing; Substance Abuse; Opioid Dependance; Inmate Population
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral counseling (Other)
  Interventions: Behavioral: Intensive Case Management

INTERVENTIONS:
Behavioral: Intensive Case Management — Transitions involves the integration of evidence-based interventions, intensive case management that incorporates outreach elements similar to assertive community treatment (ACT). Intensive case management goes beyond the tenets of case management and incorporates community outreach. This model of case management has its roots in assertive community treatment (ACT) and has demonstrated a 37% greater reduction in homelessness and a 26% greater improvement in psychiatric symptom severity compared with standard case management treatments. As such, intensive case management is likely to result in important outcomes for the target population, is evidence-based and has been validated in prison-release programs.

SUMMARY:
TRANSITIONS, a novel jail-release program for People Living with HIV/AIDS (PLWHA), will use evidence-based interventions and adapt them to create a comprehensive transitional program in Waterbury and New Haven County, Connecticut. Evidence-based interventions will include, but not be limited to, enhanced rapid HIV testing within the New Haven Community Correctional Center (NHCCC, local jail), intensive case management, continuity of buprenorphine treatment from the jail to the community setting and a novel Money Management (MM) program.

The HIV in Prisons Program and the Community Health Care Van (CHCV) at the Yale University AIDS Program, in collaboration with the Connecticut Department of Correction and the Waterbury Hospital Infectious Diseases Clinic, propose to expand the availability of opiate substitution treatment and to enhance clinical and social services for PLWHA, who are transitioning from the jail to the community setting.

As part of Transitions, we will develop a model Money Management program that we have used in community settings to improve health outcomes for socially and medically marginalized populations and adapt it for a jail-release program. The Transitions program will incorporate these elements into a combined intervention and will result in a clinical trial to compare the additional contribution of a money management program.

DETAILED DESCRIPTION:
TRANSITIONS, a novel jail-release program for People Living with HIV/AIDS (PLWHA), will use evidence-based interventions and adapt them to create a comprehensive transitional program in New Haven County, Connecticut. Evidence-based interventions will include, but not be limited to, enhanced rapid HIV testing within the New Haven Community Correctional Center (NHCCC, local jail), intensive case management, continuity of buprenorphine treatment from the jail to the community setting and a novel Money Management (MM) program that is predicated on contingency management and has been used to reduce recidivism to jail, homelessness, mental and social instability and improve social functioning. Individuals to be targeted for rapid HIV testing will be those who enter the facility with substance use disorder and mental illness. All individuals who are either diagnosed with the enhanced HIV testing or who self-identify as being HIV+ will be evaluated by the Infectious Diseases Contact Nurse (IDCN) who will work in collaboration with the Referrals Coordinator (RC). The IDCN will coordinate the medical care of the detainee within the correctional setting while the Referrals Coordinator will begin the process of coordinating the care upon release and work with the Intensive Case Managers in New Haven and Waterbury upon release.

The HIV in Prisons Program and the Community Health Care Van (CHCV) at the Yale University AIDS Program, in collaboration with the Connecticut Department of Correction and the Waterbury Hospital Infectious Diseases Clinic, propose to expand the availability of opiate substitution treatment and to enhance clinical and social services for PLWHA, who are transitioning from the jail to the community setting in New Haven county. This work builds on our previous work to enhance HIV testing in prisons and jails, , , to provide comprehensive HIV services within prisons and jails, , to implement the country's first buprenorphine treatment program in jails, to establish effective prison-released programs for sentenced prisoners, to establish buprenorphine treatment programs in mobile outreach and in HIV clinical care settings in the community, , and to establish adherence programs for PLWHA in community settings. Each of these programs and milestones have been evidence-based, rigorously studied and have resulted in replication in many parts of the country. As part of Transitions, we will develop a model Money Management program that we have used in community settings to improve health outcomes for socially and medically marginalized populations and adapt it for a jail-release program. The Transitions program will incorporate these elements into a combined intervention and will result in a clinical trial to compare the additional contribution of a money management program. The target population will include drug users who are either being released from or who have recently been released from prison or jail. Individuals will be fully assessed by a jail-based Referrals Coordinator and an intensive case manager (ICM) and a treatment plan organized. Screening and referral will take place either prior to release from the correctional setting or after release to the New Haven or Waterbury communities. HIV+ jail inmates who are returning to New Haven and Waterbury will be eligible for this study. As part of a randomized controlled trial, a subset of these will be randomized 2:1 to a Money Management program that will be adapted for our population. Direct services provided by Transitions will include enhanced rapid HIV testing within the jail setting, continuity of buprenorphine treatment from the correctional system to the community setting, intensive case management provided as modified Assertive Community Treatment and provision of a Money Management service. The strengths of this proposal are the:

* Addressing unmet medical, drug treatment, case management needs in New Haven county - these are statewide priority areas for PLWHA according to our state needs assessment;
* Collective experience and expertise in the collaboration between the Yale University HIV in Prisons Program, the CHCV, the Connecticut Department of Correction, the Waterbury Hospital ID Clinic, and a number of collaborating institutions within New Haven County;
* Novelty of introducing an approved treatment modality for opiate dependence (buprenorphine), that to date, has not been fully expanded to meet the needs of PLWHA;
* Novelty of prescribing opiate substitution therapy for released prisoners with DSM-IV criteria for opioid dependence BEFORE relapse to drug use;
* Novelty that the Connecticut Department of Correction is the first and most comprehensive system to provide buprenorphine for supervised opiate withdrawal (detox) for opioid dependent patients, thus allowing for its prescription as part of a relapse prevention program from prison and/or jail;
* Benefit of having an integrated correctional system that means that the jails and prisons are one system in Connecticut and thus able to track inmates throughout both the jail and prison system;
* Novelty of applying an evidence-based Money Manager program to released prisoners, most of whom have significant problems with substance abuse, mental illness and homelessness;
* Use of evidence-based interventions, including elements of buprenorphine maintenance treatment, intensive case management teams and money management strategies to retain released jail detainees with multiple medical and social co-morbidities.

TRANSITIONS is a novel demonstration program for managing HIV+ clients as they transition from the jail to the community setting in New Haven County, Connecticut. TRANSITIONS builds on our previous experience with developing and evaluating novel projects: 1) Project TLC (Kaiser Family Foundation, Altice, PI), the country's first transitional case management program for sentenced prisoners; 2) Project BEST (SAMHSA, Altice, PI), the country's first buprenorphine induction and stabilization program administered through a mobile health care program; and 3) and Project BELIEVE (HRSA, Altice, PI), one of ten SPNS projects integrating buprenorphine into HIV clinical care settings. Dr. Altice is also the PI for Project PLUS, two federally funded studies to develop and test pre-release (CDC, Altice, PI) and post-release (NIDA, Altice, PI) risk reduction interventions for HIV+ prisoners. The target population includes HIV+ jail detainees from New Haven County who are either being released from or who have recently been released from jail. Prison-release programs where sufficient time to plan for discharge have demonstrated significant success, however guidance for jail-release programs is urgently needed. This jail population desperately needs integrated services because of the high prevalence of HIV/AIDS, mental illness and recurrent homelessness that this incredibly vulnerable population faces as it attempts to reintegrate into the community.

Central to TRANSITIONS, we propose to develop and integrate effective, evidence-based interventions that include the following elements: 1) intensive case management (ICM) which is community-based outreach that employs feature of assertive community treatment; 2) opiate substitution therapy, primarily in the form of buprenorphine maintenance therapy; 3) enhanced communication linkages between the jail and the community. Eligible clients will include those who are HIV+ and who are either pre-release or who were released within the past 30 days. All eligible patients will receive these core elements. All Transitions clients will then be randomized 2:1 to receive additional Money Management (MM) services or no additional services. Money Management services, whose principles are predicated on contingency management, have been demonstrated to stabilize patients through improved social functioning, adherence to care, and decreased homelessness and substance misuse among patients with substance use disorder and severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

* HIV Seropositive
* 18 years of age or older
* male and female
* incarcerated but not sentenced inmates
* releasing to New Haven area
* releasing to Waterbury area
* within 30 days post release from jail

Exclusion Criteria:

Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Substance use outcomes measured by self-report | weekly reporting
Urine toxicology results | weekly report

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Clinical Research, New Haven, Connecticut
  - Waterbury Hosp ID Clinic, Waterbury, Connecticut

REFERENCES:
- [Background] Chen NE, Meyer JP, Avery AK, Draine J, Flanigan TP, Lincoln T, Spaulding AC, Springer SA, Altice FL. Adherence to HIV treatment and care among previously homeless jail detainees. AIDS Behav. 2013 Oct;17(8):2654-66. doi: 10.1007/s10461-011-0080-2. PMID 22065234
- [Background] Althoff AL, Zelenev A, Meyer JP, Fu J, Brown SE, Vagenas P, Avery AK, Cruzado-Quinones J, Spaulding AC, Altice FL. Correlates of retention in HIV care after release from jail: results from a multi-site study. AIDS Behav. 2013 Oct;17 Suppl 2(0 2):S156-70. doi: 10.1007/s10461-012-0372-1. PMID 23161210
- [Background] Chitsaz E, Meyer JP, Krishnan A, Springer SA, Marcus R, Zaller N, Jordan AO, Lincoln T, Flanigan TP, Porterfield J, Altice FL. Contribution of substance use disorders on HIV treatment outcomes and antiretroviral medication adherence among HIV-infected persons entering jail. AIDS Behav. 2013 Oct;17 Suppl 2(0 2):S118-27. doi: 10.1007/s10461-013-0506-0. PMID 23673792
- [Background] Williams CT, Kim S, Meyer J, Spaulding A, Teixeira P, Avery A, Moore K, Altice F, Murphy-Swallow D, Simon D, Wickersham J, Ouellet LJ. Gender differences in baseline health, needs at release, and predictors of care engagement among HIV-positive clients leaving jail. AIDS Behav. 2013 Oct;17 Suppl 2(0 2):S195-202. doi: 10.1007/s10461-012-0391-y. PMID 23314801
- [Background] Fu JJ, Herme M, Wickersham JA, Zelenev A, Althoff A, Zaller ND, Bazazi AR, Avery AK, Porterfield J, Jordan AO, Simon-Levine D, Lyman M, Altice FL. Understanding the revolving door: individual and structural-level predictors of recidivism among individuals with HIV leaving jail. AIDS Behav. 2013 Oct;17 Suppl 2(0 2):S145-55. doi: 10.1007/s10461-013-0590-1. PMID 24037440
- [Background] Zelenev A, Marcus R, Kopelev A, Cruzado-Quinones J, Spaulding A, Desabrais M, Lincoln T, Altice FL. Patterns of homelessness and implications for HIV health after release from jail. AIDS Behav. 2013 Oct;17 Suppl 2(0 2):S181-94. doi: 10.1007/s10461-013-0472-6. PMID 23657757
- [Background] Krishnan A, Wickersham JA, Chitsaz E, Springer SA, Jordan AO, Zaller N, Altice FL. Post-release substance abuse outcomes among HIV-infected jail detainees: results from a multisite study. AIDS Behav. 2013 Oct;17 Suppl 2(0 2):S171-80. doi: 10.1007/s10461-012-0362-3. PMID 23142854